CLINICAL TRIAL: NCT06643065
Title: The Influence of the Vaginal Microbiome on Clinical Pregnancy in Patients Undergoing a Euploid Embryo Transfer: a Prospective Blinded Multicentre Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Fundación IVI (Other)
Collaborators: Juno (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2403-JUN-096-KS
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Vaginal Microbiome
Keywords: Female reproductive tract microbiome,; Vaginal dysbiosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — vaginal swabs and blood draws
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group-1: normal microbiome
- Group-2: dysbiotic microbiome

SUMMARY:
Microorganisms such as bacteria live naturally on and in the bodies and are of great importance for our health. In the female body, almost 10% of all microorganisms live in the reproductive organs and especially in the vagina. Healthy bacteria in the vagina can defend against harmful bacteria and infections. However, it occasionally happens that the balance between healthy and harmful bacteria is disturbed, and it is believed that this could potentially harm pregnancy. However, there is not much evidence to prove a connection between an imbalance in bacteria and having an unsuccessful pregnancy.

For this reason, the goal of our study is to determine if women with certain vaginal bacteria are more likely to experience pregnancy failures. If the investigators find this to be true, patients undergoing fertility treatment might be recommended regular tests in the future. If an imbalance in bacteria is found, doctors could provide treatment to restore a healthy vaginal environment, potentially improving the chances of a successful pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* ART patients undergoing the transfer of a euploid embryo

Exclusion Criteria:

* Patients with a body mass index (BMI) ≥35

  * Patients with uncorrected uterine malformations
  * Patients with a unicornuate uterus
  * Patients with a bicornuate uterus
  * Patients with any type of submucosal myoma
  * Patients with an intramural myoma if ≥4 cm
  * Patients with severe adenomyosis (>50% of the uterine corpus affected as defined by the MUSA criteria [19])
  * Patients undergoing transfer of an embryo with a morphology score <4BC (according to the Gardner & Schoolcraft scoring system [18])
  * Patients undergoing transfer of a day-7 embryo
  * Patients who took antibiotics in the month prior to the embryo transfer (excluding antibiotics given following oocyte retrieval)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Eligible study participants are female ART patients scheduled for a frozen euploid embryo transfer
Sampling Method: Non-Probability Sample
Enrollment: 1573 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
microbial DNA extraction using molecular techniques such as qPCR | day of embryo transfer (between days 18 and 21 of the menstrual cycle)
  microbial composition. Detection (i.e., presence or absence) of the targeted bacteria and their quantification (i.e., the relative amount of each bacterial species present in the sample).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Capalbo, Study Director — JUNO GENETICS
Locations (10):
- Spain (10):
  - Ginefiv Barcelona, Barcelona, Barcelona
  - IVI Barcelona, Barcelona, Barcelona
  - IVI Bilbao, Bilbao, Bilbao
  - IVI Madrid, Madrid, Madrid
  - Ginefiv Madrid, Madrid, Madrid
  - IVI Málaga, Málaga, Málaga
  - Ginemed Sevilla, Seville, Sevilla
  - IVI Valencia, Valencia, Valencia
  - IVI Vigo, Vigo, Vigo
  - IVI Zaragoza, Zaragoza, Zaragoza